CLINICAL TRIAL: NCT00882193
Title: Pilot Therapy Using Betaine in Combination With Peginterferon Alpha-2a Plus Ribavirin in Subjects With Genotype 1 Hepatitis C Who Have Not Achieved a Sustained Viral Response With a Prior Course of Pegylated Interferon and Ribavirin
Brief Title: Pilot Study of Betaine + Combination Antiviral Therapy for Chronic Hepatitis C Genotype 1 Non-responder/Relapsers
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: new medications with improved response released
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0133-09-FB
Record Dates: First submitted 2009-04-15; First posted 2009-04-16 (Estimated); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Chronic Hepatitis C; Genotype 1; Relapse
Keywords: Chronic hepatitis C; Genotype 1; Nonresponder; Relapser; Betaine; Antiviral therapy
MeSH Terms: conditions — Hepatitis C, Chronic; Recurrence | interventions — Betaine; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Safety & Efficacy of Betaine Combined with Standard Anti-viral Therapy (Experimental): The primary objective is to examine safety & efficacy of betaine when combined with standard anti-viral therapy in previously treated adult subjects with chronic hepatitis C infected with genotype 1. Efficacy will be determined through comparison of the sustained viral response (SVR) to our protocol three-drug regimen (Betaine, Peginterferon plus Ribavirin) to that historically seen in relapsers and non-responders when retreated with standard therapy (Peginterferon and Ribavirin alone).
  Betaine (trimethylglycine) dose is 10 gm twice a day for 48 weeks. Pegasys (peginterferon alpha 2a) dose is 180mcg/0.5 ml subcutaneous injection for 48 weeks. Coegus (ribavirin) dose is 200mg - weight based, 1000 - 1200 mg/day for body weight or 75mg in 2 divided doses.
  Interventions: Drug: Betaine; Drug: Peginterferon alpha 2a; Drug: Ribavirin

INTERVENTIONS:
Drug: Betaine — Betaine 20 gm/day in 2 divided doses for 48 weeks
  Other Names: trimethylglycine
Drug: Peginterferon alpha 2a — Peginterferon alpha 2a 180mcg/0.5ml by subcutaneous injection weekly for 48 weeks
  Other Names: Pegasys
Drug: Ribavirin — Ribavirin 200mg - weight based, 1000 - 1200 mg/day for body weight < or > 75mg in 2 divided doses
  Other Names: Copegus

SUMMARY:
This is a non-randomized, open-label study examining the safety and efficacy of betaine in addition to standard anti-viral therapy in genotype 1 hepatitis C non-responders or relapsers to previous pegylated interferon plus ribavirin. Betaine (20 gm/day) in 2 divided doses will be added to Peginterferon alpha 2a (180 mcg) plus weight-based Ribavirin (1000 or 1200 mg/day, for body weight < or > 75 kg, respectively, for 48 weeks. Patients must be diagnosed with chronic hepatitis C, genotype I, and have undergone therapy for hepatitis C with pegylated interferon plus ribavirin. Subjects will be followed for safety, tolerability, hepatitis C viral response and the effect on interferon gene signaling in peripheral blood mononuclear cells during therapy.

DETAILED DESCRIPTION:
The primary objective is to examine the safety and efficacy of the betaine when combined with standard anti-viral therapy in previously treated adult subjects with chronic hepatitis C infected with genotype 1. The efficacy will be determined through comparison of the sustained viral response (SVR) to our protocol three-drug regimen (Betaine, Peginterferon plus Ribavirin) to that historically seen in relapsers and non-responders when retreated with standard therapy (Peginterferon and Ribavirin alone).

Secondary objectives include: (1) the comparison of the occurrence of rapid and early virologic response in the first 4 (Rapid Virologic Response, RVR) and 12 (Early Virologic Response, EVR) weeks of therapy, respectively, between the study regimen and historically treated patients. (2) the comparison of ALT normalization between the two groups. and (3) the effect on interferon gene signaling in peripheral blood mononuclear cells (PBMCs) between the two groups in the first 12 weeks of therapy and 6 months following the end of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be willing to give informed consent and be able to adhere to dose and visit schedules.
* History of chronic hepatitis C, genotype 1, non-responders or relapsers as documented by genotype testing and HCV RNA levels at 12 weeks ( < 2 log change) during therapy or at 3 - 12 months post therapy, respectively.
* Adult subjects 18-70 years of age, of either gender
* Liver biopsy within 3 years prior to the screening 1 visit with a pathology report confirming that the histological diagnosis is consistent with chronic hepatitis C.
* Compensated liver disease with the following maximum hematologic, biochemical and serologic criteria at the Screening visit (WNL=within normal limits) Hemoglobin > 12 g/dl for females and >13 g/dl for males, WBC > 3000/mm3, Platelets > 80,000/mm3, Direct Bilirubin - WNL. Indirect bilirubin - WNL, Albumin - WNL, Serum Creatinine - WNL.
* Fasting glucose should be 70 -140 mg/dl, results between 116-140 require a HbA1c < 8.5%
* TSH - WNL
* Subjects with a history of mild depression may be considered for entry in to this study provided that a pretreatment assessment of the subject's affective status supports that the subject is clinically stable.
* Subjects with a history of substance abuse must have abstained from using the substance for at least one year prior to the Screening visit.
* Antinuclear antibodies (ANA) < 1:320
* No radiologic evidence of a focal mass suggestive of hepatoma and/or ascites.

Exclusion Criteria:

* Pregnant or nursing subjects. Subjects who intend to become pregnant during the study period. Subjects with partners who intend to become pregnant during the study period.
* Prior response to therapy and failure to achieve SVR which may have been due to treatment non-compliance, in the assessment of the investigator based upon subject's medical history.
* Participation in any clinical trial of a HCV protease inhibitor of any duration. Subjects may have received other investigational agents for the treatment of HCV, as long as they have also received an adequate course of Peg-IFN/RBV [i.e., the investigational agent could not have replaced either Peg-IFN (such as Albuferon) or RBV (viramidine)].
* History of new hepatitis C exposure within the last 6 months
* Current or intended use of G-CSF and/or GM-CSF during the stud period is prohibited. Current use of erythropoietin (EPO) is prohibited.
* Suspected hypersensitivity to any interferon product or ribavirin
* Participation in any other clinical trial within 30 days of Screening visit 1
* Treatment with any investigational drug within 30 days of Screening visit 1.
* Any other cause for liver disease other than CHC, including but not limited to: hemachromatosis, Alpha-1 antitrypsin deficiency, Wilson's disease, Autoimmune hepatitis, Alcoholic liver disease, Non-alcoholic steatohepatitis (NASH), Drug-related liver disease
* Known coagulopathies including hemophilia
* Known hemoglobinopathies
* Known G6PD deficiency
* Known coinfection with HIV and/or HBV
* Evidence of active or suspected malignancy or a history of malignancy within the last five years (with the exception of adequately treated basal cell carcinoma of the skin).
* Evidence of decompensated liver disease such as history or presence of ascites, bleeding varices or hepatic encephalopathy
* Subjects with organ transplants other than cornea or hair transplant
* Any Known preexisting medical condition, that could interfere with the subject's participation in and completion of the study including, but not limited to moderate to severe depression, or a history of severe psychiatric disorder, such as psychosis, suicidal ideation and/or suicidal attempt; Subjects with a past history or current use of lithium and/or antipsychotic drugs; CNS trauma or seizure disorder; Clinically significant ECG abnormalities and/or significant cardiovascular dysfunction within the past 2 years prior to Screening ; Poorly controlled diabetes mellitis; Chronic pulmonary disease (COPD); Immunologically mediated disease such as inflammatory bowel disease, rheumatoid arthritis, idiopathic thrombocytopenia purpura, systemic lupus erythematosus, autoimmune hemolytic anemia, scleroderma, severe psoriasis or symptomatic thyroid disorder; Any medical condition requiring, or likely to require during the course of the study, chronic systemic administration of steroids: History of, or active clinical gout.
* Substance abuse, such as alcohol (>80 g/day), IV drugs and inhaled drugs. Subjects with a history of substance abuse must have abstained from the abuse substance for at least one year. Subjects with clinically significant retinal abnormalities
* Any other condition which in the opinion of the investigator would make the subject unsuitable for enrollment, or could interfere with the subject participating in and completing the protocol
* Subjects who are part of the staff personnel directly involved with the study
* Subjects who are immediate family members of the investigational study staff

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2009-05-01 (Actual); Primary Completion 2011-01-12 (Actual); Study Completion 2011-01-12 (Actual)

PRIMARY OUTCOMES:
Safety and efficacy of betaine combined with standard antiviral therapy | 72 weeks
  To examine the safety and efficacy of betaine when combined with standard antiviral therapy in previously treated subjects with chronic hepatitis c genotype 1

SECONDARY OUTCOMES:
Effect on interferon gene signaling in peripheral blood mononuclear cells | 72 weeks
  The effect on interferon gene signaling in peripheral blood mononuclear cells in the first 12 weeks of treatment and 6 months following the end of therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Mark E Mailliard, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States